CLINICAL TRIAL: NCT00005150
Title: Minnesota Heart Health Program
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1021; R01HL025523 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Myocardial Infarction; Hypertension; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Stroke; Myocardial Infarction; Hypertension; Coronary Disease

SUMMARY:
To conduct a large-scale community-based demonstration and education research project designed to evaluate the effectiveness of multiple educational strategies on risk factor reduction and the primary prevention of population-wide cardiovascular diseases in three intervention communities compared with three control communities. The program was evaluated by cross-sectional surveys, a longitudinal survey, and morbidity and mortality surveillance.

DETAILED DESCRIPTION:
BACKGROUND:

The rationale for prevention derives from the mass nature of adult cardiovascular diseases in affluent societies, the insidious development of the underlying processes, particularly hypertension and atherosclerosis, the high immediate out-of hospital mortality of coronary disease and stroke, and the long-term excessive risk after survival of an initial episode.

The potential for a preventive approach in cardiovascular diseases was based on the large differences in disease rates found between populations and the strong associations between individual risk factor levels and disease rates within high risk cultures. The congruence of these population observations with clinical evidence and with plausible mechanisms of cause, strengthened inference of their causal importance. Further, the safety and feasibility were well established of modifying individuals' cardiovascular risk characteristics and changing personal health behavior through medical and educational strategies. Finally, the dynamic nature of the changes in vital statistics on deaths reported from hypertension, stroke, and coronary heart disease (CHD) in many nations, at the rate of one to two percent a year and greater, both upward and downward, indicated their preventability, though none of these trends was adequately explained when the study began in 1980.

The rationale for a population or community-wide strategy, as in the Minnesota Heart Health Program, contrasted to a high-risk individual, medical approach, was based on all the above considerations, plus the demonstration that entire populations were at excess risk relative to others. Focusing solely on the portion of higher risk people among high risk cultures appeared to be a necessary medical part of a community-wide prevention approach, but it was insufficient and inefficient as a sole or major public health strategy. This was mainly because the bulk of attributable (excess) cases of cardiovascular disease came from the large central part of the population distribution of risk, not the tail. The socially learned behaviors which lead to the precursors of cardiovascular disease were also mass phenomena, requiring a population strategy of prevention and health promotion. Finally, concentration of preventive effort only among the high risk or only on adults tended to ignore the mass emergence of youth into early adulthood bearing the physical characteristics of excess risk and already having well-developed unhealthy behaviors. Therefore, a rational and effective public health strategy would appear to be one directed toward all ages and segments of the community, over a sustained period, with the ultimate objective to prevent elevated risk and risky behaviors in the first place.

DESIGN NARRATIVE:

Three pairs of communities were selected, each pair with one education and one control community. Communities were matched on size and distance from Minneapolis-St. Paul and pairs were similar in median income, education, health care, and media resources. The first pair, Mankato and Winona, were small agricultural communities of approximately 40,000 in population in 1980. The second pair, Fargo, North Dakota and Moorhead, Minnesota paired with Sioux Falls, South Dakota, were medium-sized urban centers of approximately 100,000 in population. Bloomington and Roseville, Minnesota were suburban centers in the Twin Cities metropolitan area with a population of approximately 80,000.

The education program began in Mankato in 1981 after two baseline surveys, in Fargo-Moorhead in 1982 after three baseline surveys, and in Bloomington in 1983 after four baseline surveys. Education activities continued in the three communities for five years concluding in the staged manner in which they began. Targeted risk factors included blood pressure, exercise habits, smoking, and blood cholesterol levels. Health messages were communicated by involvement of community leaders and organizations, media education, population-based risk factor screening and education, adult education classes, youth and parent education disseminated in schools, health professional's educa0tion, and community-wide risk factor education campaigns.

The effectiveness of the program was evaluated by annual population survey samples of cross-sections or cohorts and by morbidity and mortality surveillance. The annual risk factor survey measured community and individual change in risk factors and related behaviors in 25-74 year old persons living in each of the six sites. Annual surveys included between 300-500 persons and were population-based, random, neighborhood cluster samples of each town. Selected households were invited to participate. A home interview was conducted to collect data on health beliefs, attitudes, and behaviors, medical history, health message exposure, and demographic characterization. After the home interview, participants had additional risk factor measurements at a survey center. Data were collected on height, weight, blood pressure, serum total and HDL cholesterol, and serum thiocyanate. In each community, a 50 percent sample of subjects was assessed for dietary habits and the other 50 percent for physical activity.

Morbidity and mortality data on myocardial infarction and stroke were collected and analyzed for the Minnesota Heart Health Program areas and mortality data for all of Minnesota, North Dakota, and South Dakota. Computer classification algorithms were developed jointly with the Pawtucket Heart Health Program and the Stanford Five-City Multifactor Risk Reduction Program to allow pooling of data of the three studies. All hospitalized cases of myocardial infarction and stroke were investigated and cause of death was validated for cardiovascular disease deaths occurring out-of-hospital. Deaths occurring throughout Minnesota, North and South Dakota were catalogued. Hospital disease surveillance was carried out with the cooperation of 34 area hospitals. Mortality was ascertained by death certificate counts and from tapes supplied by the three State Health Departments. Morbidity and mortality data were compared between pooled education versus pooled comparison communities and mortality data were compared between these and the remaining areas of the three states.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1980-07; Study Completion 1993-06

REFERENCES:
- [Background] Murray DM, Perry CL, Davis MA: Cardiovascular Risk Reduction in Children. Education and Treatment of Children, 10(1):48-57, 1987
- [Background] Perry CL, Crockett SJ, Pirie P: Influencing Parental Health Behavior: Implications of Community Assessments. Health Educ, 18:5, 1987
- [Background] Perry CL, Klepp KI, Halper A, Dudovitz B, Golden D, Griffin G, Smyth M: Promoting Healthy Eating and Physical Activity Patterns Among Adolescents: A Pilot Study of 'Slice of Life' Health Educ Research, 2(2):93-103, 1987
- [Background] Perry CL, Silvis GL. Smoking prevention: behavioral prescriptions for the pediatrician. Pediatrics. 1987 May;79(5):790-9. PMID 3575039
- [Background] Sorensen G, Pechacek TF. Attitudes toward smoking cessation among men and women. J Behav Med. 1987 Apr;10(2):129-37. doi: 10.1007/BF00846421. PMID 3612774
- [Background] Perry CL, Murray DM, Klepp KI; Centers for Disease Control (CDC). Predictors of adolescent smoking and implications for prevention. MMWR Suppl. 1987 Sep 4;36(4):41S-45S. No abstract available. PMID 3116396
- [Background] Jeffery RW: Behavioral Treatment of Obesity. Ann Behav Med, 9(1):20-24, 1987
- [Background] Jeffery RW, Forster JL: Obesity as a Public Health Problem, Chapter 11. In: Johnson WG (Ed), Advances in Eating Disorders, Vol. I: Treating and Preventing Obesity. Greenwich, CT: Jai Press, Inc., pp 253-271, 1987
- [Background] Silvis GL, Perry CL. Understanding and deterring tobacco use among adolescents. Pediatr Clin North Am. 1987 Apr;34(2):363-79. doi: 10.1016/s0031-3955(16)36221-6. PMID 3550658
- [Background] Jeffery RW. Dietary risk factors and their modification in cardiovascular disease. J Consult Clin Psychol. 1988 Jun;56(3):350-7. doi: 10.1037//0022-006x.56.3.350. No abstract available. PMID 3294260
- [Background] Perry CL. Results of prevention programs with adolescents. Drug Alcohol Depend. 1987 Sep;20(1):13-9. doi: 10.1016/0376-8716(87)90071-8. PMID 3678039
- [Background] Bracht NF. Use of community analysis methods in community-wide intervention programs. Scand J Prim Health Care Suppl. 1988;1:23-30. PMID 3227199
- [Background] Rastam L, Luepker RV, Mittelmark MB, Murray DM, Slater JS, Blackburn H. Population screening and referral for hypercholesterolemia. Am J Prev Med. 1988 Sep-Oct;4(5):249-54. PMID 3224001
- [Background] Rastam L, Admire JB, Frantz ID Jr, Hellerstedt W, Hunninghake DM, Kuba K, Luepker RV. Measurement of blood cholesterol with the Reflotron analyzer evaluated. Clin Chem. 1988 Feb;34(2):426. No abstract available. PMID 3342525
- [Background] Mittelmark MB, Leupker RV, Grimm R Jr, Kottke TE, Blackburn H. The role of physicians in a community-wide program for prevention of cardiovascular disease: the Minnesota Heart Health Program. Public Health Rep. 1988 Jul-Aug;103(4):360-5. PMID 3136495
- [Background] Murray DM, Kurth CL, Finnegan JR Jr, Pirie PL, Admire JB, Luepker RV. Direct mail as a prompt for follow-up care among persons at risk for hypertension. Am J Prev Med. 1988 Nov-Dec;4(6):331-5. PMID 3228529
- [Background] Rastam L, Luepker RV, Pirie PL. Effect of screening and referral on follow-up and treatment of high blood cholesterol levels. Am J Prev Med. 1988 Sep-Oct;4(5):244-8. PMID 3224000
- [Background] Forster JL, Jeffery RW, Snell MK. One-year follow-up study to a worksite weight control program. Prev Med. 1988 Jan;17(1):129-33. doi: 10.1016/0091-7435(88)90078-3. PMID 3362799
- [Background] Crockett SJ, Mullis RM, Perry CL. Parent nutrition education: a conceptual model. J Sch Health. 1988 Feb;58(2):53-7. doi: 10.1111/j.1746-1561.1988.tb05822.x. PMID 3352225
- [Background] Jeffery RW, Pheley AM, Forster JL, Kramer FM, Snell MK. Payroll contracting for smoking cessation: a worksite pilot study. Am J Prev Med. 1988 Mar-Apr;4(2):83-6. PMID 3395495
- [Background] Mullis RM, Pirie P. Lean meats make the grade--a collaborative nutrition intervention program. J Am Diet Assoc. 1988 Feb;88(2):191-5. PMID 3339206
- [Background] Perry CL, Klepp KI, Shultz JM. Primary prevention of cardiovascular disease: communitywide strategies for youth. J Consult Clin Psychol. 1988 Jun;56(3):358-64. doi: 10.1037//0022-006x.56.3.358. No abstract available. PMID 3294261
- [Background] Perry CL, Luepker RV, Murray DM, Kurth C, Mullis R, Crockett S, Jacobs DR Jr. Parent involvement with children's health promotion: the Minnesota Home Team. Am J Public Health. 1988 Sep;78(9):1156-60. doi: 10.2105/ajph.78.9.1156. PMID 3407811
- [Background] Forster JL, Jeffery RW, Schmid TL, Kramer FM. Preventing weight gain in adults: a pound of prevention. Health Psychol. 1988;7(6):515-25. doi: 10.1037//0278-6133.7.6.515. PMID 3215160
- [Background] Glanz K, Mullis RM. Environmental interventions to promote healthy eating: a review of models, programs, and evidence. Health Educ Q. 1988 Winter;15(4):395-415. doi: 10.1177/109019818801500403. PMID 3068206
- [Background] Luepker RV, Perry CL, Murray DM, Mullis R. Hypertension prevention through nutrition education in youth: a school-based program involving parents. Health Psychol. 1988;7 Suppl:233-45. PMID 3243221
- [Background] Blake SM, Klepp KI, Pechacek TF, Folsom AR, Luepker RV, Jacobs DR, Mittelmark MB. Differences in smoking cessation strategies between men and women. Addict Behav. 1989;14(4):409-18. doi: 10.1016/0306-4603(89)90028-2. PMID 2789466
- [Background] Jeffery RW, Forster JL, Folsom AR, Luepker RV, Jacobs DR Jr, Blackburn H. The relationship between social status and body mass index in the Minnesota Heart Health Program. Int J Obes. 1989;13(1):59-67. PMID 2703294
- [Background] Crockett SJ, Mullis R, Perry CL, Luepker RV. Parent education in youth-directed nutrition interventions. Prev Med. 1989 Jul;18(4):475-91. doi: 10.1016/0091-7435(89)90007-8. PMID 2678093
- [Background] Perry CL, Luepker RV, Murray DM, Hearn MD, Halper A, Dudovitz B, Maile MC, Smyth M. Parent involvement with children's health promotion: a one-year follow-up of the Minnesota home team. Health Educ Q. 1989 Summer;16(2):171-80. doi: 10.1177/109019818901600203. PMID 2732061
- [Background] Sorensen G, Pechacek TF. Implementing nonsmoking policies in the private sector and assessing their effects. N Y State J Med. 1989 Jan;89(1):11-5. PMID 2784199
- [Background] Finnegan JR Jr, Murray DM, Kurth C, McCarthy P. Measuring and tracking education program implementation: the Minnesota Heart Health Program experience. Health Educ Q. 1989 Spring;16(1):77-90. doi: 10.1177/109019818901600109. PMID 2703350
- [Background] Lando HA, Loken B, Howard-Pitney B, Pechacek T. Community impact of a localized smoking cessation contest. Am J Public Health. 1990 May;80(5):601-3. doi: 10.2105/ajph.80.5.601. PMID 2109545
- [Background] Mullis R, Shannon B. Building partnerships with the food marketing system: an expanding role for dietitians. J Am Diet Assoc. 1987 Dec;87(12):1632-4. No abstract available. PMID 3680820
- [Background] Weisbrod RR, Pirie PL, Bracht NF. Impact of a community health promotion program on existing organizations: the Minnesota Heart Health Program. Soc Sci Med. 1992 Mar;34(6):639-48. doi: 10.1016/0277-9536(92)90191-r. PMID 1574731
- [Background] Weisbrod RR, Bracht NF, Pirie PL, Veblen-Mortenson S. Current status of health promotion activities in four midwest cities. Public Health Rep. 1991 May-Jun;106(3):310-7. PMID 1905053
- [Background] Weisbrod RR, Pirie PL, Bracht NF, Elstun P. Worksite health promotion in four Midwest cities. J Community Health. 1991 Jun;16(3):169-77. doi: 10.1007/BF01323975. PMID 1860969
- [Background] Rastam L, Hannan PJ, Luepker RV, Mittelmark MB, Murray DM, Slater JS. Seasonal variation in plasma cholesterol distributions: implications for screening and referral. Am J Prev Med. 1992 Nov-Dec;8(6):360-6. PMID 1482576
- [Background] Arneson T, Luepker R, Pirie P, Sinaiko A. Cholesterol screening by primary care pediatricians: a study of attitudes and practices in the Minneapolis-St Paul metropolitan area. Pediatrics. 1992 Mar;89(3):502-5. PMID 1741228
- [Background] Luepker RV, Perry CL. The Minnesota Heart Health Program. Education for youth and parents. Ann N Y Acad Sci. 1991;623:314-21. doi: 10.1111/j.1749-6632.1991.tb43740.x. PMID 2042839
- [Background] Bostick RM, Luepker RV, Kofron PM, Pirie PL. Changes in physician practice for the prevention of cardiovascular disease. Arch Intern Med. 1991 Mar;151(3):478-84. PMID 2001129
- [Background] Lichtenstein E, Lando HA, Nothwehr F. Readiness to quit as a predictor of smoking changes in the Minnesota Heart Health Program. Health Psychol. 1994 Sep;13(5):393-6. doi: 10.1037//0278-6133.13.5.393. PMID 7805633
- [Background] Troein M, Arneson T, Rastam L, Pirie PL, Selander S, Luepker RV. Reported treatment of hypercholesterolemia by family physicians in Sweden and Minnesota. Am J Prev Med. 1995 Sep-Oct;11(5):324-8. PMID 8573363
- [Background] Troein M, Arneson T, Rastam L, Pirie PL, Selander S, Luepker RV. Reported treatment of hypertension by family physicians in Sweden and Minnesota: a physician survey of practice habits. J Intern Med. 1995 Sep;238(3):215-21. doi: 10.1111/j.1365-2796.1995.tb00925.x. PMID 7673850
- [Background] Jeffery RW, Gray CW, French SA, Hellerstedt WL, Murray D, Luepker RV, Blackburn H. Evaluation of weight reduction in a community intervention for cardiovascular disease risk: changes in body mass index in the Minnesota Heart Health Program. Int J Obes Relat Metab Disord. 1995 Jan;19(1):30-9. PMID 7719388
- [Background] Luepker RV, Murray DM, Jacobs DR Jr, Mittelmark MB, Bracht N, Carlaw R, Crow R, Elmer P, Finnegan J, Folsom AR, et al. Community education for cardiovascular disease prevention: risk factor changes in the Minnesota Heart Health Program. Am J Public Health. 1994 Sep;84(9):1383-93. doi: 10.2105/ajph.84.9.1383. PMID 8092360
- [Background] Strickland D, Sprafka JM, Luepker RV, Grimm RH Jr. Association of antihypertensive agents and blood lipids in a population-based survey. Epidemiology. 1994 Jan;5(1):96-101. doi: 10.1097/00001648-199401000-00014. PMID 8117788
- [Background] Blackburn H: The Public Health View of Diet and Mass Hyperlipidemia. Part I, Part II. Cardiovas Rev Rep, 1:361-369, 433-442, 1980
- [Background] Blackburn H, Gillum RF: Heart Disease. In: Public Health and Preventive Medicine, 11th Edition, Last JM (Ed), Appleton-Century-Crofts, New York, pp 1168-1201, 1980
- [Background] Pechacek TF: Strategies for the Modification of Smoking Behavior: A Synoptic Review. Behavioral Medicine Update, 1:16-18, 1980
- [Background] Pechacek TF, McAlister A: Strategies for the Modification of Smoking Behavior: Treatment and Prevention. In: A Comprehensive Handbook of Behavioral Medicine, Ferguson J, Taylor B (Eds), Spectrum Publications, New York, pp 257-298, 1980
- [Background] Prineas RJ, Gillum RF, Blackburn H: Possibilities for Primary Prevention of Hypertension. In: Childhood Prevention of Atherosclerosis and Hypertension, Lauer RM, Shekelle RB (Eds), Raven Press, New York, pp 357-366, 1980
- [Background] Luepker RV, Pechacek TF, Murray DM, Johnson CA, Hund F, Jacobs DR. Saliva thiocyanate: a chemical indicator of cigarette smoking in adolescents. Am J Public Health. 1981 Dec;71(12):1320-4. doi: 10.2105/ajph.71.12.1320. PMID 7315995
- [Background] Arkin RM, Roemhild HF, Johnson CA, Luepker RV, Murray DM. The Minnesota smoking prevention program: a seventh-grade health curriculum supplement. J Sch Health. 1981 Nov;51(9):611-6. doi: 10.1111/j.1746-1561.1981.tb02246.x. PMID 6913699
- [Background] Blackburn H: A Public Health Approach to Diet, Risk Factors and Coronary Heart Disease. In: Hyperlipidemia (A Cornell Postgraduate Course), Scheidt S (Ed), MedCom Inc., New York, pp 27-35, 1981
- [Background] Blackburn H: Primary Prevention of Coronary Heart Disease. In: Clinical Medicine, Spittell J Jr. (Ed), Harper & Row, Philadelphia, pp 1-23, 1981
- [Background] Pirie P, Jacobs D, Jeffery R, Hannan P. Distortion in self-reported height and weight data. J Am Diet Assoc. 1981 Jun;78(6):601-6. PMID 7252014
- [Background] Coates TJ, Jeffery RW, Slinkard LA. Heart healthy eating and exercise: introducing and maintaining changes in health behaviors. Am J Public Health. 1981 Jan;71(1):15-23. doi: 10.2105/ajph.71.1.15. PMID 7258426
- [Background] Prevention of coronary heart disease. World Health Organ Tech Rep Ser. 1982;678:1-53. No abstract available. PMID 6812294
- [Background] Carlaw RW, DiAngelis NM. Promoting health and preventing disease some thoughts for HMOs. Health Educ Q. 1982 Spring;9(1):81-95. doi: 10.1177/109019818200900106. PMID 7076509
- [Background] Coates TJ, Petersen A, Perry C (Eds): Promoting Adolescent Health: A Dialog on Research and Practice. Academic Press, New York, 1982
- [Background] Gatewood L: Evaluation of Prognostic Indices After Acute MI. Proceedings of Scientific Meeting on Ischemic Heart Disease, Specialized Centers of Research, NHLBI, Bethesda, MD, May 1982
- [Background] Grimm RH Jr, Luepker RV, Taylor H, Blackburn H. Long-term effects of a blood pressure survey on patient treatment in a community. Circulation. 1982 May;65(5):946-50. doi: 10.1161/01.cir.65.5.946. PMID 7074758
- [Background] Jeffery RW, Pirie PL, Rosenthal BS, Gerber WM, Murray DM. Nutrition education in supermarkets: an unsuccessful attempt to influence knowledge and product sales. J Behav Med. 1982 Jun;5(2):189-200. doi: 10.1007/BF00844808. PMID 7131542
- [Background] Leon A, Blackburn H: Physical Activity and Hypertension. In: Hypertension. Cardiology I, Sleight P, Freis E (Eds), Butterworths, London, pp 14-36, 1982
- [Background] Loken B. Heavy smokers', light smokers', and nonsmokers' beliefs about cigarette smoking. J Appl Psychol. 1982 Oct;67(5):616-22. No abstract available. PMID 7142102
- [Background] Mittelmark MB, Murray DM, Luepker RV, Pechacek TF. Cigarette smoking among adolescents: is the rate declining? Prev Med. 1982 Nov;11(6):708-12. doi: 10.1016/0091-7435(82)90032-9. No abstract available. PMID 7163146
- [Background] Perry C: Adolescent Health: An Education-Ecological Perspective. In: Promoting Adolescent Health: A Dialog on Research and Practice. Coates T, Petersen A, Perry C (Eds), Academic Press, New York, pp 73-86, 1982
- [Background] Blackburn H: Determinants of Individual and Population Blood Lipoprotein Levels: Nutritional-Genetic Interactions. In: Genetic Factors in Nutrition, Velasquez A, Gourges H (Eds), Academic Press, New York, 1983
- [Background] Blackburn H. Diet and atherosclerosis: epidemiologic evidence and public health implications. Prev Med. 1983 Jan;12(1):2-10. doi: 10.1016/0091-7435(83)90161-5. No abstract available. PMID 6844305
- [Background] Blackburn H: Physical Activity and Coronary Heart Disease: A Brief Update and Population View. Parts I, II. J Cardiac Rehab, 3:101-111, 171-174, 1983
- [Background] Blackburn H. Research and demonstration projects in community cardiovascular disease prevention. J Public Health Policy. 1983 Dec;4(4):398-421. No abstract available. PMID 6662913
- [Background] Blackburn H, Prineas R. Diet and hypertension: anthropology, epidemiology, and public health implications. Prog Biochem Pharmacol. 1983;19:31-79. No abstract available. PMID 6338525
- [Background] DiAngelis N, Luepker RV. The effect of the dental setting on blood pressure measurement. Am J Public Health. 1983 Oct;73(10):1210-2. doi: 10.2105/ajph.73.10.1210. PMID 6614279
- [Background] Ettema JS, Brown JW, Luepker RV. Knowledge gap effects in a health information campaign. Public Opin Q. 1983 Winter;47(4):516-27. doi: 10.1086/268809. PMID 10264839
- [Background] Folsom AR, Kuba K, Leupker RV, Jacobs DR, Frantz ID Jr. Lipid concentrations in serum and EDTA-treated plasma from fasting and nonfasting normal persons, with particular regard to high-density lipoprotein cholesterol. Clin Chem. 1983 Mar;29(3):505-8. PMID 6402325
- [Background] Gillum RF, Prineas RJ, Jeffery RW, Jacobs DR, Elmer PJ, Gomez O, Blackburn H. Nonpharmacologic therapy of hypertension: the independent effects of weight reduction and sodium restriction in overweight borderline hypertensive patients. Am Heart J. 1983 Jan;105(1):128-33. doi: 10.1016/0002-8703(83)90289-2. No abstract available. PMID 6849226
- [Background] Jacobs DR Jr, Anderson JT, Hannan P, Keys A, Blackburn H. Variability in individual serum cholesterol response to change in diet. Arteriosclerosis. 1983 Jul-Aug;3(4):349-56. doi: 10.1161/01.atv.3.4.349. PMID 6882289
- [Background] Perry CL, Murray DM. Enhancing the transition years: the challenge of adolescent health promotion. J Sch Health. 1982 May;52(5):307-11. doi: 10.1111/j.1746-1561.1982.tb04628.x. No abstract available. PMID 6919708
- [Background] Jeffery RW, Gillum R, Gerber WM, Jacobs D, Elmer PJ, Prineas RJ. Weight and sodium reduction for the prevention of hypertension: a comparison of group treatment and individual counseling. Am J Public Health. 1983 Jun;73(6):691-3. doi: 10.2105/ajph.73.6.691. PMID 6846677
- [Background] Kline FG: The Minnesota Heart Health Project: Field Intervention in American Communities. In: Att Forandra Levnadssatt: Rapport fran ett Symposium om Metoder att Forbattra Folkhalsan (In: To Change Lifestyles: Report From a Symposium on Methods to Improve Public Health). Arvidsson O (Ed), Riksbankens Jubileumsfond, Stockholm, 1983
- [Background] Kottke TE, Foels JK, Hill C, Choi T, Fenderson DA. Perceived palatability of the prudent diet: results of a dietary demonstration for physicians. Prev Med. 1983 Jul;12(4):588-94. doi: 10.1016/0091-7435(83)90211-6. PMID 6622440
- [Background] Leon A, Blackburn H: Physical Inactivity. In: Prevention of Coronary Heart Disease, Kaplan NM, Stamler J (Ed), W.B. Saunders Co., New York, pp 86-97, 1983
- [Background] Luepker RV, Johnson CA, Murray DM, Pechacek TF. Prevention of cigarette smoking: three-year follow-up of an education program for youth. J Behav Med. 1983 Mar;6(1):53-62. doi: 10.1007/BF00845276. PMID 6687341
- [Background] McKee D: The Effects of Family and Public Health Education on Preventive Health Behavior. The Case of Changes in Smoking, Exercise and Dietary Behavior. Doctoral Dissertation, Department of Family Social Science, University of Minnesota, Minneapolis, 1983
- [Background] Mullis R: Health Promotion Opportunities. Community Nutritionist, January-February, pp 11-12, 1983
- [Background] Pavlik JV: The Effects of Two Health Information Campaigns on the Complexity of Cognitive Structure: An Information Processing Approach. Doctoral Dissertation, School of Journalism, University of Minnesota, Minneapolis, 1983
- [Background] Pechacek TF, Grimm RH: Cigarette Smoking and the Prevention of Coronary Disease: Principles for Effective Smoking Cessation Programs for Health Professionals. In: Physician's Guide to the Prevention of Coronary Heart Disease. Podell RN, Stewart MM (Eds), Addison-Wesley, Palo Alto, pp 34-77, 1983
- [Background] Prineas RJ, Jacobs D. Quality of Korotkoff sounds: bell vs diaphragm, cubital fossa vs brachial artery. Prev Med. 1983 Sep;12(5):715-9. doi: 10.1016/0091-7435(83)90229-3. PMID 6657637
- [Background] Sopko G, Jacobs DR Jr, Jeffery R, Mittelmark M, Lenz K, Hedding E, Lipchik R, Gerber W. Effects on blood lipids and body weight in high risk men of a practical exercise program. Atherosclerosis. 1983 Dec;49(3):219-29. doi: 10.1016/0021-9150(83)90134-x. PMID 6581808
- [Background] Pirie PL, Luepker RV, Jacobs DR Jr, Brown JW, Hall N. Development and validation of a self-scoring test for coronary heart disease risk. J Community Health. 1983 Fall;9(1):65-79. doi: 10.1007/BF01318934. PMID 6678259
- [Background] Blackburn H, Luepker R, Kline FG, Bracht N, Carlaw R, Jacobs DR, Mittelmark M, Stauffer L, Taylor HL: The Minnesota Heart Health Program: A Research and Demonstration Project in Cardiovascular Disease Prevention. In: Behavioral Health: A Handbook for Health Enhancement and Disease Prevention, Matarazzo J et al (Eds), John Wiley & Sons, New York, 1984
- [Background] Jeffery RW, Pirie PL, Elmer PJ, Bjornson-Benson WM, Mullenbach VA, Kurth CL, Johnson SL. Low-sodium, high-potassium diet: feasibility and acceptability in a normotensive population. Am J Public Health. 1984 May;74(5):492-4. doi: 10.2105/ajph.74.5.492. PMID 6711725
- [Background] Pechacek TF, Fox BH, Murray DM, Luepker RV: Review of Techniques for Measurement of Smoking. In: Behavioral Health: A Handbook of Health Enhancement and Disease Prevention. Matarazzo J, et al (Eds) John Wiley & Sons, New York, 1984
- [Background] Folsom AR, Pechacek TF, de Gaudemaris R, Luepker RV, Jacobs DR Jr, Gillum RF. Consumption of 'low-yield' cigarettes: its frequency and relationship to serum thiocyanate. Am J Public Health. 1984 Jun;74(6):564-8. doi: 10.2105/ajph.74.6.564. PMID 6426329
- [Background] Folsom AR, Prineas RJ, Jacobs DR, Luepker RV, Gillum RF. Measured differences between fourth and fifth phase diastolic blood pressures in 4885 adults: implications for blood pressure surveys. Int J Epidemiol. 1984 Dec;13(4):436-41. doi: 10.1093/ije/13.4.436. PMID 6519881
- [Background] Kottke TE, Foels JK, Hill C, Choi T, Fenderson DA. Nutrition counseling in private practice: attitudes and activities of family physicians. Prev Med. 1984 Mar;13(2):219-25. doi: 10.1016/0091-7435(84)90053-7. PMID 6330723
- [Background] Luepker RV, Jacobs DR, Brown JW, Sobel JL, Prineas R. Hypertension control in two rural communities. Minn Med. 1984 Jun;67(6):341-4. No abstract available. PMID 6472236
- [Background] Mullis RM, Bowen PE. Process guides for nutrition care in community health. J Am Diet Assoc. 1985 Jan;85(1):73-6. PMID 3965545
- [Background] Perry CL. A conceptual approach to school-based health promotion. J Sch Health. 1984;54(6):33-8. PMID 6565118
- [Background] Sopko G, Jacobs DR Jr, Taylor HL. Dietary measures of physical activity. Am J Epidemiol. 1984 Dec;120(6):900-11. doi: 10.1093/oxfordjournals.aje.a113961. PMID 6507429
- [Background] Carlaw RW, Mittlemark MB, Bracht N, Luepker R. Organization for a community cardiovascular health program: experiences from the Minnesota Heart Health Program. Health Educ Q. 1984 Fall;11(3):243-52. doi: 10.1177/109019818401100303. PMID 6520005
- [Background] Blackburn H, Pechacek T: Smoking Cessation and the Minnesota Heart Health Program. In: Proceedings of the 5th World Conference on Smoking and Health, Nosbakken D (Ed), 1984
- [Background] Glasgow RE, Klesges RC, Mizes JS, Pechacek TF. Quitting smoking: strategies used and variables associated with success in a stop-smoking contest. J Consult Clin Psychol. 1985 Dec;53(6):905-12. doi: 10.1037//0022-006x.53.6.905. No abstract available. PMID 4086690
- [Background] Perry CL, Mullis RM, Maile MC. Modifying the eating behavior of young children. J Sch Health. 1985 Dec;55(10):399-402. doi: 10.1111/j.1746-1561.1985.tb01163.x. PMID 3853032
- [Background] Perry CL, Griffin G, Murray DM. Assessing needs for youth health promotion. Prev Med. 1985 May;14(3):379-93. doi: 10.1016/0091-7435(85)90064-7. PMID 4059190
- [Background] Mittelmark MB, Luepker RV, Jacobs DR, Bracht NF, Carlaw RW, Crow RS, Finnegan J, Grimm RH, Jeffery RW, Kline FG, et al. Community-wide prevention of cardiovascular disease: education strategies of the Minnesota Heart Health Program. Prev Med. 1986 Jan;15(1):1-17. doi: 10.1016/0091-7435(86)90031-9. PMID 3714655
- [Background] Mullis RM, Lansing D: Using Focus Groups to Plan Worksite Nutrition Programs. J Nutr Educ, Special Supplement, 18(2):32-33, 1986
- [Background] Perry CL, Klepp KI, Halper A, Hawkins KG, Murray DM. A process evaluation study of peer leaders in health education. J Sch Health. 1986 Feb;56(2):62-7. doi: 10.1111/j.1746-1561.1986.tb01176.x. PMID 3633365
- [Background] Pirie PL, Elias WS, Wackman DB, Jacobs DR Jr, Murray DM, Mittelmark MB, Luepker RV, Blackburn H. Characteristics of participants and nonparticipants in a community cardiovascular disease risk factor screening: the Minnesota Heart Health Program. Am J Prev Med. 1986 Jan-Feb;2(1):20-5. PMID 3453156
- [Background] Sorensen G, Pechacek T, Pallonen U. Occupational and worksite norms and attitudes about smoking cessation. Am J Public Health. 1986 May;76(5):544-9. doi: 10.2105/ajph.76.5.544. PMID 3963283
- [Background] Crow R, Blackburn H, Jacobs D, Hannan P, Pirie P, Mittelmark M, Murray D, Luepker R. Population strategies to enhance physical activity: the Minnesota Heart Health Program. Acta Med Scand Suppl. 1986;711:93-112. doi: 10.1111/j.0954-6820.1986.tb08937.x. PMID 3465209
- [Background] Folsom AR, Jacobs DR Jr, Caspersen CJ, Gomez-Marin O, Knudsen J. Test-retest reliability of the Minnesota Leisure Time Physical Activity Questionnaire. J Chronic Dis. 1986;39(7):505-11. doi: 10.1016/0021-9681(86)90195-5. PMID 3722314
- [Background] Murray DM, Luepker RV, Pirie PL, Grimm RH Jr, Bloom E, Davis MA, Blackburn H. Systematic risk factor screening and education: a community-wide approach to prevention of coronary heart disease. Prev Med. 1986 Nov;15(6):661-72. doi: 10.1016/0091-7435(86)90071-x. PMID 3797397
- [Background] Murray DM. Dissemination of community health promotion programs: the Fargo-Moorhead Heart Health Program. J Sch Health. 1986 Nov;56(9):375-81. doi: 10.1111/j.1746-1561.1986.tb05776.x. PMID 3640927
- [Background] Jacobs DR Jr, Luepker RV, Mittelmark MB, Folsom AR, Pirie PL, Mascioli SR, Hannan PJ, Pechacek TF, Bracht NF, Carlaw RW, et al. Community-wide prevention strategies: evaluation design of the Minnesota Heart Health Program. J Chronic Dis. 1986;39(10):775-88. doi: 10.1016/0021-9681(86)90080-9. PMID 3760106
- [Background] Venters M, Jacobs DR Jr, Pirie P, Luepker RV, Folsom AR, Gillum RF. Marital status and cardiovascular risk: the Minnesota Heart Survey and the Minnesota Heart Health Program. Prev Med. 1986 Nov;15(6):591-605. doi: 10.1016/0091-7435(86)90064-2. PMID 3797391
- [Background] Salonen JT, Kottke TE, Jacobs DR Jr, Hannan PJ. Analysis of community-based cardiovascular disease prevention studies--evaluation issues in the North Karelia Project and the Minnesota Heart Health Program. Int J Epidemiol. 1986 Jun;15(2):176-82. doi: 10.1093/ije/15.2.176. PMID 3721679
- [Background] Luepker R, Murray D, Prineas R. [Primary prevention of hypertension in childhood (the population approach)]. Kardiologiia. 1986 Jan;26(1):69-77. Russian. PMID 3951137
- [Background] Mullis RM, Perry CL, Pirie PL: A Model for Levels of Community Health Promotion. In: Coates AY and Frankle RT (Eds), Nutrition in the Community: The Art of Delivering Services, 2nd Edition. St. Louis: Times Mirror/Mosby College Publishing, 1986
- [Background] Murray D, Luepker R, Grimm R, Blackburn H. [Prevention and treatment of hypertension at the population level: the Minnesota Heart Health Program]. Kardiologiia. 1986 Jan;26(1):78-84. Russian. PMID 3951138
- [Background] Blackburn H: Atherosclerosis and Coronary Heart Disease. Strategy for Change: A Population Approach to Prevention. In: Fidge NH, Nestel PJ (Eds), Atherosclerosis VII. New York: Elsevier Science Publishers B.V., pp 15-17, 1986
- [Background] Murray DM, Leupker RV, Grimm R, Blackburn H: Prevention and Treatment of Hypertension at a Community Level: The Minnesota Heart Health Program. In: Horan MJ, Shkvatsabaya IK (Eds), Hypertension: Psychophysiological, Biobehavioral, and Epidemiological Aspects. NIH Publication No. 86-2704, Washington, DC: U.S. Government Printing Office, pp 183-191, 1986
- [Background] Luepker RV, Murray DM, Prineas RJ: Primary Prevention of Hypertension in Youth: A Population Approach. In: Horan MJ, Shkvatsabaya IK (Eds), Hypertension: Psychophysiological, Biobehavioral, and Epidemiological Aspects. NIH Publication No. 86-2704, Washington, DC: U.S. Government Printing Office, pp 211-226, 1986
- [Background] Luepker RV: Coronary Heart Disease Risk Factor Reduction in the Elderly. Quality of Life and Cardiovascular Care, 2(4):159-175, 1986
- [Background] Luepker RV: Prevention of Cigarette Smoking. In: Feldman DA, Stiffman AR (Eds), Advances in Adolescent Mental Health. Greenwich, CT: JAI Press, Inc, 1986
- [Background] Forster JL, Bloom E, Sorensen G, Jeffery RW, Prineas RJ. Reproductive history and body mass index in black and white women. Prev Med. 1986 Nov;15(6):685-91. doi: 10.1016/0091-7435(86)90073-3. PMID 3797399
- [Background] Perry CL. Community-wide health promotion and drug abuse prevention. J Sch Health. 1986 Nov;56(9):359-63. doi: 10.1111/j.1746-1561.1986.tb05772.x. PMID 3640925
- [Background] Sorensen G, Pechacek T. Occupational and sex differences in smoking and smoking cessation. J Occup Med. 1986 May;28(5):360-4. PMID 3486965
- [Background] Blake SM, Jeffery RW, Finnegan JR, Crow RS, Pirie PL, Ringhofer KR, Fruetel JR, Caspersen CJ, Mittelmark MB: Process Evaluation of a Community-Based Physical Activity Campaign: The Minnesota Heart Health Program Experience. Health Educ Research, 2(2):115-121, 1987
- [Background] Finnegan JR, Loken B, Howard-Pitney B: Using Direct Mail to Bridge 'Knowledge Gaps' in Communication About Health. J Direct Marketing, 1(Summer):3, 1987
- [Background] Loken B, Pirie PL, Virnig K, Hinkle R, Salmon CT: The Use of 0-10 Scales in Telephone Surveys. J Market Res Society, 29(3):353-362, 1987
- [Background] Mullis RM, Hunt MK, Foster M, Hachfeld L, Lansing D, Synder P, Pirie P: Environmental Support of Healthful Food Behavior: The Shop Smart For Your Heart Grocery Program. J Nutr Educ, 19(5):225-228, 1987